CLINICAL TRIAL: NCT03826030
Title: TRANScranial Direct Current Stimulation for POst-stroke Motor Recovery - a Phase II sTudy (TRANSPORT 2)
Brief Title: Transcranial Direct Current Stimulation for Post-stroke Motor Recovery
Acronym: TRANSPORT 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00103316; U01NS102353 (NIH)
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Stroke, Ischemic; Motor Activity; Upper Extremity Paralysis
Keywords: stroke; stroke recovery; brain stimulation; transcranial direct current stimulation
MeSH Terms: conditions — Ischemic Stroke; Motor Activity; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Sham tDCS + mCIMT (Sham Comparator): Sham tDCS (Transcranial direct current stimulation) administers no dose or zero milliampere stimulation through the tDCS device, during Constraint Induced Movement Therapy (mCIMT)
  Interventions: Device: Sham; Behavioral: mCIMT
- 2 mA tDCS + mCIMT (Active Comparator): 2 mA tDCS (Transcranial direct current stimulation) administers low dose or 2 milliampere stimulation through the tDCS device, during Constraint Induced Movement Therapy (mCIMT)
  Interventions: Device: Low dose tDCS; Behavioral: mCIMT
- 4 mA + mCIMT (Active Comparator): 4 mA tDCS (Transcranial direct current stimulation) administers high dose or 4 milliampere stimulation through the tDCS device, during Constraint Induced Movement Therapy (mCIMT)
  Interventions: Device: High dose tDCS; Behavioral: mCIMT

INTERVENTIONS:
Device: Sham — Sham group only receives 30 seconds of stimulation at 2mA in the beginning to create a sensory perception to the scalp in order to blind the subject.
  Arms: Sham tDCS + mCIMT
Device: Low dose tDCS — The low dose tDCS group receives direct current stimulation at 2 mA for 30 minutes per session
  Arms: 2 mA tDCS + mCIMT
Device: High dose tDCS — The high dose tDCS group receives direct current stimulation at 4 mA for 30 minutes per session
  Arms: 4 mA + mCIMT
Behavioral: mCIMT — All three tDCS groups receive constraint-induced movement therapy as the adjunctive behavioral therapy for 2 hours per session

SUMMARY:
This research study is to find out if brain stimulation at different dosage level combined with an efficacy-proven rehabilitation therapy can improve arm function. The stimulation technique is called transcranial direct current stimulation (tDCS). The treatment uses direct currents to stimulate specific parts of the brain affected by stroke. The adjunctive rehabilitation therapy is called "modified Constraint-Induced Movement Therapy" (mCIMT). During this therapy the subject will wear a mitt on the hand of the arm that was not affected by a stroke and force to use the weak arm. The study will test 3 different doses of brain stimulation in combination with mCIMT to find out the most promising one.

ELIGIBILITY:
Each subject must meet all of the following criteria to participate in this study:

1. 18-80 years old; and
2. First-ever unihemispheric ischemic stroke radiologically verified and occurred within the past 30-180 days; and
3. >10° of active wrist extension, >10° of thumb abduction/extension, and > 10° of extension in at least 2 additional digits; and
4. Unilateral limb weakness with a Fugl-Meyer Upper Extremity score of ≤ 54 (out of 66) to avoid ceiling effects; and
5. An absolute difference of FM-UE scores between the two baseline assessments that is ≤ 2 points indicating stable motor impairment; if subject is not stable, then he/she will be invited for a reassessment after 7-14 days (but no more than 3 reassessments); and
6. Pre-stroke mRS ≤2; and
7. Signed informed consent by the subject or Legally Authorized Representative (LAR).

Each Subject who meets any of the following criteria will be excluded from the study:

1. Primary intracerebral hematoma, subarachnoid hemorrhage or bi-hemispheric or bilateral brainstem ischemic strokes;
2. Medication use at the time of study that may interfere with tDCS, including but not limited to carbamazepine, flunarizine, sulpiride, rivastigmine, dextromethorphan;
3. Other co-existent neuromuscular disorders (pre- or post-stroke) affecting upper extremity motor function;
4. Other neurological disorders (pre- or post-stroke) affecting subject's ability to participate in the study;
5. Moderate to severe cognitive impairment defined as Montreal Cognitive Assessment (MOCA) score < 18/30;
6. History of medically uncontrolled depression or other neuro-psychiatric disorders despite medications either before or after stroke that may affect subject's ability to participate in the study;
7. Uncontrolled hypertension despite medical treatment(s) at the time of randomization, defined as SBP≥185 mmHg or DBP≥110 mmHg (patient can be treated, reassessed and randomized later);
8. Presence of any MRI/tDCS/TMS risk factors including but not limited to: 8a) an electrically, magnetically or mechanically activated metallic or nonmetallic implant including cardiac pacemaker, intracerebral vascular clips or any other electrically sensitive support system; 8b) a non-fixed metallic part in any part of the body, including a previous metallic injury to eye; 8c) pregnancy (effects of MRI, TMS, and tDCS on the fetus are unknown); 8d) history of seizure disorder or post-stroke seizure; 8e) preexisting scalp lesion under the intended electrode placement or a bone defect or hemicraniectomy;
9. Planning to move from the local area within the next 6 months;
10. Life expectancy less than 6 months;
11. Has received Botulinum toxin injection to the affected upper extremity in the past 3 months prior to randomization or expectation that Botulinum will be given to the Upper Extremity prior to the completion of the last follow-up visit;
12. Concurrent enrollment in another investigational stroke recovery study;
13. Doesn't speak sufficient English to comply with study procedures;
14. Expectation that subject cannot comply with study procedures and visits.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Feng, MD, Principal Investigator — Duke University; Gottfried Schlaug, MD, PhD, Principal Investigator — Baystate Health
Locations (14):
- United States (14):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - Keck Hospital of USC, Los Angeles, California
  - MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia
  - Emory Rehabilitation Hospital, Atlanta, Georgia
  - Cardinal Hill Rehabilitation Hospital, Lexington, Kentucky
  - Baystate Medical Center, Springfield, Massachusetts
  - Burke Rehabilitation Center, White Plains, New York
  - Duke University Hospital, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland VA Medical Center, Cleveland, Ohio
  - Moss Rehabilitation Research Institute, Elkins Park, Pennsylvania
  - University of Pittsburgh Medical Center Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina University Hospital, Charleston, South Carolina
  - Memorial Hermann Texas Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
We will follow the National Institute of Health Stroke Trial Network policy and procedure to share IPD. Please refer to https://nihstrokenet.org/ for detailed information.
Time Frame: Please refer to https://nihstrokenet.org/ for detailed information in term of time-frame of sharing such data
Access Criteria: Please refer to https://nihstrokenet.org/ for detailed information in term of time-frame of sharing such data
URL: https://nihstrokenet.org/

REFERENCES:
- [Derived] Schlaug G, Cassarly C, Feld JA, Wolf SL, Rowe VT, Fritz S, Chhatbar PY, Shinde A, Su Z, Broderick JP, Zorowitz R, Awosika O, Edwards D, Lin C, Franciso GE, Wittenberg GF, Pundik S, Gregory C, Borich MR, Ramakrishnan V, Feng W. Safety and efficacy of transcranial direct current stimulation in addition to constraint-induced movement therapy for post-stroke motor recovery (TRANSPORT2): a phase 2, multicentre, randomised, sham-controlled triple-blind trial. Lancet Neurol. 2025 May;24(5):400-412. doi: 10.1016/S1474-4422(25)00044-4. Epub 2025 Mar 26. PMID 40157380

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham tDCS + mCIMT: Sham tDCS + mCIMT group only receives 30 seconds of stimulation at 2mA in the beginning to create a sensory perception to the scalp in order to blind the subject. All three tDCS groups receive constraint-induced movement therapy as the adjunctive behavioral therapy for 2 hours per session.
- 2 mA tDCS + mCIMT: 2 mA tDCS + mCIMT group receives direct current stimulation at 2 mA for 30 minutes per session. All three tDCS groups receive constraint-induced movement therapy as the adjunctive behavioral therapy for 2 hours per session.
- 4 mA + mCIMT: 4 mA tDCS + mCIMT group receives direct current stimulation at 4 mA for 30 minutes per session. All three tDCS groups receive constraint-induced movement therapy as the adjunctive behavioral therapy for 2 hours per session.
Period: Overall Study
Arm/Group | Sham tDCS + mCIMT | 2 mA tDCS + mCIMT | 4 mA + mCIMT
Started | 43 | 43 | 43
Completed | 39 | 42 | 41
Not Completed | 4 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Too busy to return for visits | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham tDCS + mCIMT | 2 mA tDCS + mCIMT | 4 mA + mCIMT | Total
Number analyzed (Participants) | 43 | 43 | 43 | 129
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56.0 [46.0 to 66.0] | 62.0 [51.0 to 67.0] | 60.0 [51.0 to 67.0] | 59.0 [50.0 to 66.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 13 | 19 | 54
  Male | 21 | 30 | 24 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 5 | 11
  Not Hispanic or Latino | 40 | 40 | 38 | 118
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 20 | 14 | 19 | 53
  White | 23 | 25 | 21 | 69
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 2 | 2
Time from Index Stroke to Randomization [Count of Participants; unit: Participants]
  30-90 Days | 11 | 12 | 11 | 34
  91-180 Days | 32 | 31 | 32 | 95
Pre-Stroke Dominant Side [Count of Participants; unit: Participants]
  Left | 3 | 4 | 3 | 10
  Right | 40 | 39 | 40 | 119
Side of the Body Made Weak by the Index Stroke [Count of Participants; unit: Participants]
  Left | 23 | 30 | 17 | 70
  Right | 20 | 13 | 26 | 59
Pre-Stroke Modified Rankin Scale (mRS) [Count of Participants; unit: Participants] — The MRS has a score range of 0 to 6, where a higher score indicates poorer function.
  Participants
    0: No Symptoms At All | 39 | 35 | 35 | 109
    1: No Significant Disability Despite Symptoms | 1 | 4 | 5 | 10
    2: Slight Disability | 3 | 4 | 3 | 10
Fugl-Meyer Upper-Extremity (FM-UE) Scale [Median (Inter-Quartile Range); unit: units on a scale] — The Fugl-Meyer Upper-Extremity (FM-UE) is a measure of motor impairment (0 to 66 points, with higher points indicating less impairment). FM-UE scale consists of a 33-item assessment which provides a global assessment of UE motor impairment.
  units on a scale | 39.0 [30.0 to 46.0] | 39.0 [27.0 to 48.0] | 40.0 [27.0 to 48.0] | 39.0 [27.0 to 47.0]
Montreal Cognitive Assessment (MoCA) [Median (Inter-Quartile Range); unit: units on a scale] — The MoCA has a score range of 0 to 30, where a higher score indicates better cognitive function.
  units on a scale | 27.0 [25.0 to 29.0] | 27.0 [24.0 to 29.0] | 26.0 [23.0 to 28.0] | 27.0 [24.0 to 28.0]
NIH Stroke Scale (NIHSS) [Median (Inter-Quartile Range); unit: units on a scale] — The NIHSS has a score range of 0 to 42, where a higher score indicates greater stroke severity.
  units on a scale | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0]
Wolf-Motor Functional Test (WMFT) Time Score [Median (Inter-Quartile Range); unit: seconds] — The Wolf Motor Function Test (WMFT) is a measure of functional motor activity that quantifies upper extremity (UE) motor ability through timed and functional tasks. The WMFT Time Score the median of 15 timed arm movements and hand dexterity tasks, each to be completed in 120s. If a task could not be completed in 120s, a score of 121s was assigned. A lower WMFT Time Score is better.
  seconds | 3.9 [2.4 to 11.8] | 4.0 [2.1 to 22.2] | 3.3 [2.3 to 11.5] | 3.8 [2.3 to 12.2]
Log(WMFT Time Score) [Median (Inter-Quartile Range); unit: log(seconds)] — Logarithmic transformation of WMFT Time Score
  log(seconds) | 1.4 [0.9 to 2.5] | 1.4 [0.7 to 3.1] | 1.2 [0.8 to 2.4] | 1.3 [0.8 to 2.5]
Stroke Impact Scale (SIS) Hand Subscale [Median (Inter-Quartile Range); unit: units on a scale] — The SIS has a score range of 0 to 100, where a higher score indicates better quality of life after a stroke.
  units on a scale | 25.0 [10.0 to 30.0] | 30.0 [15.0 to 55.0] | 30.0 [15.0 to 40.0] | 25.0 [15.0 to 40.0]
Lesion Volume - Affected Side (Centrally Assessed) [Median (Inter-Quartile Range); unit: centimeters cubed] — Population: Missing for one participant randomized to Sham tDCS + mCIMT
  centimeters cubed
    number analyzed (Participants) | 42 | 43 | 43 | 128
    (all) | 1.4 [0.8 to 15.8] | 2.5 [1.2 to 12.4] | 1.5 [0.9 to 11.8] | 1.9 [0.9 to 12.1]
Weighted Corticospinal Tract (wCST) Lesion Load - Affected Side (Centrally Assessed) [Median (Inter-Quartile Range); unit: centimeters cubed] — Population: Missing for one subject randomized to Sham tDCS + mCIMT
  centimeters cubed
    number analyzed (Participants) | 42 | 43 | 43 | 128
    (all) | 0.5 [0.3 to 0.7] | 0.5 [0.3 to 0.8] | 0.6 [0.2 to 0.8] | 0.5 [0.3 to 0.8]
Presumed Motor Evoked Potential (MEP) Positive - Affected Side [Count of Participants; unit: Participants] — MEP was presumed positive if the %MSO<100 for the more affected side rMT by local TMS rater Population: Missing for one subject randomized to Sham tDCS + mCIMT.
  Participants
    number analyzed (Participants) | 42 | 43 | 43 | 128
    Yes | 32 | 31 | 27 | 90
    No | 10 | 12 | 16 | 38

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in FM-UE From Baseline
Description: The Fugl-Meyer Upper-Extremity (FM-UE) is a measure of motor impairment (0 to 66 points, with higher points indicating less impairment). FM-UE scale consists of a 33-item assessment which provides a global assessment of UE motor impairment. A rater provides an ordinal rating (2=near normal ability/response, 1=partial ability, 0=unable to perform/no response). The FM-UE scale is a proven scale with excellent intra-rater reliability (0.99), inter-rater reliability (0.99), test-retest reliability (0.94 -0.99), and internal consistency (0.97). FM-UE scale was assessed both by site raters (who were masked to the intervention) and by a central rater (who was masked to timepoint and intervention), by watching video recordings. The centrally rated score was used for the primary outcome analysis. For each element of the FM-UE scale, if the centrally rated score could not be determined, the site rater score was substituted.
Time Frame: Day 15
Population: Modified intent to treat population which included all subjects with any post-baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sham tDCS + mCIMT | 2 mA tDCS + mCIMT | 4 mA + mCIMT
Number analyzed (Participants) | 41 | 43 | 43
units on a scale | 4.91 [3.00 to 6.82] | 3.87 [2.00 to 5.74] | 5.53 [3.64 to 7.42]
Statistical Analysis 1: Comparison: Sham tDCS + mCIMT vs 2 mA tDCS + mCIMT vs 4 mA + mCIMT; The null hypothesis was no overall difference in FM-UE scale change between the three groups on day 15. The change in FM-UE was modelled using a linear mixed-effects repeated measures model adjusted for visit (ie, day 15, day 45, and day 105), treatment group, treatment group by visit interaction, baseline FM-UE, time from stroke (30-90 vs. 91-180 days), and enrolment site. An AR(1) autocorrelation structure was used for visit, and variance components structure for sites; Test type: Superiority; p = 0.39, Mixed Models Analysis

2. Secondary Outcome: Mean Change in WMFT Time Score From Baseline
Description: The Wolf Motor Function Test (WMFT) is a measure of functional motor activity that quantifies upper extremity (UE) motor ability through timed and functional tasks. The WMFT Time Score the median of 15 timed arm movements and hand dexterity tasks, each to be completed in 120s. If a task could not be completed in 120s, a score of 121s was assigned. A lower WMFT Time Score is better.
Time Frame: Day 15
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sham tDCS + mCIMT | 2 mA tDCS + mCIMT | 4 mA + mCIMT
Number analyzed (Participants) | 41 | 43 | 43
score on a scale | -8.67 [-15.50 to -1.84] | -1.65 [-8.76 to 5.46] | -10.37 [-18.64 to -2.11]

3. Secondary Outcome: Mean Change in SIS Hand Subscale From Baseline
Description: The Stroke Impact Scale (SIS) has 8 subscales which ask questions regarding a patient's physical limitations, memory and thinking, emotions and mood, ability to communicate, daily activities, mobility at home and in the community, use of hand most affected by stroke, and ability to participate in meaningful life activities. Each subscale item is rated on a scale from 5-1 (5= None of the time, 4=a little of the time, 3=Some of the time, 2=Most of the time, 1=All of the time). The domain/subscale scores, including the SIS Hand Subscale, range from 0 (worst) to 100 (best).
Time Frame: Day 15
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sham tDCS + mCIMT | 2 mA tDCS + mCIMT | 4 mA + mCIMT
Number analyzed (Participants) | 41 | 43 | 43
score on a scale | 25.24 [19.13 to 31.36] | 13.60 [8.01 to 19.20] | 21.51 [15.77 to 27.25]

ADVERSE EVENTS:
Time Frame: Up to 105 days after randomization
Description: Reportable adverse events (AE) included: all serious AEs, any AEs that occur during the intervention period, any AEs that are possibly or definitely related to the intervention regardless of when they occur, and all clinically important adverse safety events including: severe headache, second-degree skin burn, clinical seizure, and neurological deterioration (greater than or equal to 4 point increase in NIHSS).
Arm/Group | Sham tDCS + mCIMT | 2 mA tDCS + mCIMT | 4 mA + mCIMT
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 2/43 | 0/43 | 5/43
Other Adverse Events (participants affected / at risk) | 4/43 | 1/43 | 5/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham tDCS + mCIMT (N=43) | 2 mA tDCS + mCIMT (N=43) | 4 mA + mCIMT (N=43)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham tDCS + mCIMT (N=43) | 2 mA tDCS + mCIMT (N=43) | 4 mA + mCIMT (N=43)
Fatigue (General disorders) | 1 (3) | 1 (1) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT03826030/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT03826030/ICF_000.pdf